CLINICAL TRIAL: NCT04604444
Title: Evaluating the Effects of Intensive Speech and Language Rehabilitation Regarding Neuroplasticity, Speech, Language, Communication Skills and Quality of Life for People With Acquired Aphasia and/or Apraxia of Speech in the Chronic Phase
Brief Title: Changes in Neuroplasticity Following Intensive Rehabilitation of Aphasia and/or Apraxia of Speech
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Malaga (Other)
Responsible Party: Principal Investigator, Ellika Schalling, Professor, Speech Language Pathologist, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1651-31
Record Dates: First submitted 2020-09-11; First posted 2020-10-27 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Aphasia; Apraxia of Speech; Dysarthria
Keywords: Intensive Aphasia Rehabilitation; Intensive Apraxia of Speech Rehabilitation; Neuroplasticity
MeSH Terms: conditions — Aphasia; Apraxias; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal Intensive Rehabilitation of Aphasia/AOS (MIRAA) (Experimental): A minimum of 3 hour speech-language training daily during 10 days.
  Interventions: Behavioral: Multimodal Intensive Rehabilitation of Aphasia and Apraxia of Speech

INTERVENTIONS:
Behavioral: Multimodal Intensive Rehabilitation of Aphasia and Apraxia of Speech — Intensive Comprehensive Aphasia (ICAP) and Apraxia of Speech Program

SUMMARY:
The present study aims to investigate the short- and long-term effects of two weeks of intensive speech-language pathology intervention with additional physiotherapy, on aphasia and apraxia of speech (AOS) and their neural correlates in thirty persons with chronic stroke. Changes are studied following intensive treatment of aphasia and AOS with standardised speech-language testing and testing of communication and with voxel-based morphometry (VBM) analysis and resting state functional connectivity (rsFC).

DETAILED DESCRIPTION:
This study explores structural and functional brain changes in relation to effects on speech, language, communication and quality of life following an intensive speech-language program with additional physiotherapy for persons with chronic aphasia and/or apraxia of speech. The participants are consecutively recruited from a rehabilitation centre providing intensive treatment for chronic conditions following stroke or other neurological injuries. The speech-language pathologists (SLPs) involved in the rehabilitation programs perform the testing directly before and after intensive intervention with an additional follow up after 16 weeks (+-2) with testing of speech-language, communication and quality of life. The SLPs have more than five years of experience of working with aphasia and are specialised in working with intensive treatment, they have acquired in-depth knowledge on how to evaluate and treat aphasia and apraxia of speech in lectures and workshops. The test procedure is recorded with camcorder and voice recorder to provide the opportunity to access data retrospectively and to minimize bias by including an external SLP who makes a second blinded evaluation on randomized participants' performance in ASRS, BNT and CAT by studying the video and voice material. Structural and functional neuroplasticity is also investigated with voxel-based morphometry (VBM) analysis, resting state functional connectivity (rsFC) in domain-specific (language processing) and domain-general (executive and attention processing). This intensive neuro-rehabilitation program for speech and language deficits named Multimodal Intensive Rehabilitation for Aphasia and Apraxia of Speech (MIRAA) is defined as an ICAP (Intensive Comprehensive Aphasia Program) with focus on both speech and language function and communicative activity and participation. The program is intensive: consisting of ten days of training (5 hours/day), with a minimum of three hours dedicated to speech and language rehabilitation with additional physical therapy. The program includes both individual treatment, group therapy and computer-based therapy. The therapy is individually set up after the participant's goals together with the team including SLPs, physiotherapists and a board-certified neurologist and/or specialist in rehabilitation medicine. The goals are set by the participants, family members and clinicians the first day of the program. The participant and their significant other are offered education with the aim to enhance the knowledge on communication, the key concepts of neuroplasticity and other functions and strategies important in everyday life. The treatment methods being used are evidence-based and/or widely used multimodal programs covering the need for extensive training programs targeting both impairment-based therapy and functional communication. The specific questions are: Does ten days of with an intensive comprehensive aphasia/AOS program result in any clinical significant improvements in speech and/or language function and other cognitive skills for participants with chronic aphasia and/or apraxia of speech? Does the intensive intervention have any effect on the quality of everyday life concerning speech and language functions, activity and communicative participation for people with chronic aphasia and apraxia of speech? Can functional and anatomical brain changes be detected following ten days of intensive speech and language intervention for these participants?

ELIGIBILITY:
Inclusion Criteria:

* Aphasia 7 months post stroke diagnosed by SLP
* Apraxia of Speech 7 months post stroke diagnosed by SLP

Exclusion Criteria:

* Dementia
* Severe loss of sight
* Severe loss of hearing
* Metal implants (preventing fMRI)
* Claustrophobia (preventing fMRI)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Aphasia Test (CAT) language battery, in pilot Swedish test A-ning. | Changes from baseline in language battery scores at 2 and 18 weeks.
  Comprehension of spoken language: minimum score 0, maximum score 66; Comprehension of written langugage: minimum score 0, maximum score 62; Repetition: minimum score 0, maximum score 74; Naming: minimum score 0, maximum score no limit; Reading: minimum score 0, maximum score 70; Writing: minimum score 0, maximum score 76. Higher scores mean better outcome in language functions.
Rating scale for apraxia of speech (SkaFTA, Swedish version of ASRS) | Changes from baseline scores at 2 and 18 weeks.
  Minimum score 0, maximum score 52. Lower scores mean better outcome in speech functions.
Communication Outcome After Stroke (COAST) | Changes from baseline scores at 2 and 18 weeks.
  Minimum score 0, maximum score 100. Higher scores mean better outcome in communication.
Goal Attainment Scaling (GAS), International Classification of Functioning, Disability and Health (ICF). Aphasia adapted GAS scales for self-evaluation of communication functions, participation and activity. | Changes from baseline at week 18.
  Minimum score -2, maximum score +2. Higher scores mean better outcome in quality of life.

SECONDARY OUTCOMES:
Barrow Neurological Institute Screening for Higher Cerebral Function (BNIS) | Changes from baseline at week 2
  Minimum score 0, maximum score 50. Higher scores mean better outcome in cognition.
Boston Naming Test (BNT) | Changes from baseline at week 2 and week 18.
  Minimum score 0, maximum score 60. Higher scores mean better outcome in naming ability.
Protocol for Apraxia of Speech (TAX) | Changes from baseline at week 2 and week 18.
  Minimum score 0, maximum score 30. Lower scores mean mean better outcome in speech functions and non verbal oral apraxia.
Comprehensive Aphasia Test (CAT), subtest cognitive screening | Changes from baseline in Comprehensive Aphasia Test cognitive screening scores at 2 and 18 weeks.
  Minimum score 0, maximum score 38. Higher scores mean better outcome in cognitive functions.

CONTACTS AND LOCATIONS:
Overall Officials: Ellika Schalling, Professor, Principal Investigator — Uppsala University
Locations (1):
- Uppsala Universitet, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 2020-2030
Access Criteria: Swedish National Data Service open source http://snd.gu.se/sv/dashboard/data-description/0a1f0ee0-454e-4d66-b43f-b235bfe821a6#publications

DOCUMENTS (3):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT04604444/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT04604444/SAP_000.pdf
  • Informed Consent Form (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT04604444/ICF_001.pdf